CLINICAL TRIAL: NCT05649163
Title: A Non-interventional, Multi-cohort, Multi-center, Prospective Real-world Study of Treatment Pattern and Clinical Outcomes in Patients With HER2-overexpressed Advanced Solid Tumors After Progression of First-line Standard Therapy
Brief Title: Real-world Study of HER2-overexpressed Advanced Solid Tumors After Progression of First-line Standard Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shen Lin (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Shen Lin, Principal Investigator, Peking University
Organization: Peking University (Other)
Other Study IDs: DVReal-001
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: HER2; Advanced Gastric Cancer; Advanced Gastroesophageal Junction Adenocarcinoma; Advanced Solid Tumor
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort1: Cohort1: About 186 patients with histologically or cytologically confirmed gastric/gastroesophageal junction (GEJ) adenocarcinoma with HER2 overexpression who received a regimen containing Disitamab Vedotin;
  Interventions: Drug: Disitamab Vedotin
- Cohort2: Cohort2: About 80 patients with histologically or cytologically confirmed HER2-overexpressed gastric cancer /GEJ adenocarcinoma who received an investigator-selected regimen in addition to Disitamab Vedotin;
  Interventions: Drug: Disitamab Vedotin
- Cohort3: Cohort3: Approximately 40 patients with other advanced solid tumors histologically or cytologically confirmed with HER2-overexpression and receiving a regimen containing Disitamab Vedotin.
  Interventions: Drug: Disitamab Vedotin

INTERVENTIONS:
Drug: Disitamab Vedotin — Cohort 1: received a regimen containing Disitamab Vedotin. Cohort 2: received an investigator-selected regimen in addition to Disitamab Vedotin; Treatment options selected by the investigator: no treatment containing Disitamab Vedotin was given, and other systemic antitumor agents (including chemotherapy, such as paclitaxel, docetaxel, irinotecan, and fluorouracil) were selected by the investigator in line with clinical practice. Targeted therapy: such as apatinib, ramucirumab; Combination therapy: ramucirumab + paclitaxel; Immune checkpoint inhibitors such as PD1/PD-L1); Cohort 3: receiving a regimen containing Disitamab Vedotin.
  Other Names: RC48

SUMMARY:
The goal of this observational study is to learn about in describe treatment pattern and clinical outcomes in patients with HER2-overexpressed advanced solid tumors after progression of first-line standard therapy. The main questions it aims to answer are:

* To evaluate the real-world safety and efficacy of Disitamab Vedotin in second-line and beyond treatment of advanced solid tumors with HER2 overexpression
* To describe the treatment pattern and clinical outcomes of patients with advanced gastric cancer with HER2 overexpression in real world Settings after the failure of first-line standard therapy.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multi-cohort, multi-center real-world study to evaluate the treatment pattern and clinical outcomes of patients with advanced HER2-overexpressed solid tumors after the progression of first-line standard therapy. Enrolled subjects in this study were treated according to the treatment protocol established by physicians according to clinical routine. The tests, examinations and drug use in the study were consistent with the requirements of the clinical practice. No additional tests, examinations and drugs were generated from the data collection in this study. The study included 306 patients with HER2-overexpressed advanced gastric/gastroesophageal junction (GEJ) adenocarcinoma and other advanced solid tumors who had failed previous first-line standard therapy. HER2 overexpression was defined as IHC2+ or IHC3+ detected by immunohistochemistry (IHC) (either primary or metastatic tumor tissue).

ELIGIBILITY:
Inclusion Criteria:

* Signing informed consent and agreeing to comply with study requirements;
* Age ≥18 years old, gender unlimited;
* ECOG physical status 0-2 points;
* Patients with locally advanced or metastatic solid tumors confirmed histologically or cytologically;Cohort1-2 cohort: patients who had received at least previous first-line standard therapy (HER2 IHC3+ or IHC2+/FISH+ patients with first-line trastuzumab (or its biosimilar) combined with chemotherapy (fluorouracil and/or platinum-based chemotherapy);IHC2+/FISH- patients with first-line Immunotherapy combined with chemotherapy (fluorouracil and/or platinum-based chemotherapy) or chemotherapy alone);In Cohort3 cohort, patients received at least the standard first-line treatment clearly recommended by the guidelines. Patients with clear disease progression confirmed by the investigator or documented history.
* HER2 overexpression was defined as 2+ or 3+ immunohistochemistry (both primary and metastatic tumor tissue were acceptable), and previous patient test results (confirmed by the investigator) or center test results were acceptable.
* Have measurable or evaluable lesions according to RECIST1.1 criteria;
* The investigator evaluated that the patients would benefit from the study treatment;
* Good compliance, willing and able to follow the trial and follow-up procedures;
* Have traceable patient medical records.

Exclusion Criteria:

* Known hypersensitivity or delayed allergic reactions to certain components of the study drug or similar drugs;
* Participating in any interventional clinical trials;
* The investigator assessed inappropriate inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced solid tumors with HER2 overexpression after previous first-line standard therapy failure
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 3 and above adverse events associated with Disitamab Vedotin treatment during the study period. | From January 2023 to January 2025
  The incidence of grade 3 and above adverse events associated with Disitamab Vedotin treatment during the study period.

SECONDARY OUTCOMES:
Incidence, drug correlation, and severity of adverse events during the study period | From January 2023 to January 2025
  Incidence, drug correlation, and severity of adverse events during the study period
Overall survival (OS) | From January 2023 to January 2025
  Time from the start of administration to death from any cause
Progression-free survival (PFS) | From January 2023 to January 2025
  The first objective record of disease progression or death from any cause (whichever occurs first) occurred after patients were enrolled and given the drug
Objective response rate (ORR) | From January 2023 to January 2025
  Refers to the proportion of patients with an optimal overall response rating of CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China